CLINICAL TRIAL: NCT02102230
Title: The Impact of CBT-I on Cannabis Cessation Outcomes
Brief Title: CBT-I for Cannabis Use
Acronym: CBT-I-CU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principle Investigator as left government service
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN-016-13F
Record Dates: First submitted 2014-03-25; First posted 2014-04-02 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Marijuana Abuse; Sleep Initiation and Maintenance Disorders
Keywords: Sleep Initiation and Maintenance Disorders; marijuana abuse; Veterans
MeSH Terms: conditions — Marijuana Abuse; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Desensitization, Immunologic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CBT-I (Experimental): Group Cognitive-Behavioral Therapy for Insomnia (CBT-I)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- CBT-I-MA (Active Comparator): Group Cognitive-Behavioral Therapy for Insomnia Plus Mobile App (CBT-I-MA)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia Plus Mobile App (CBT-I-MA)
- PC (Placebo Comparator): Desensitization Treatment for Insomnia (DTI)
  Interventions: Behavioral: Desensitization Treatment for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — This is a group-delivered version of the six-session Cognitive-Behavioral Treatment for Insomnia that has been disseminated throughout the VA. It incorporates psychoeducation, diary-based sleep assessment, estimation of sleep scheduling and efficiency, evaluation/mitigation of dysfunctional sleep-related beliefs/ behaviors, generation of sleep prescription (typically restriction), iterative review of sleep efficiency and prescription, and planning for maintenance of gains.
  Other Names: CBT-I
  Arms: CBT-I
Behavioral: Cognitive Behavioral Therapy for Insomnia Plus Mobile App (CBT-I-MA) — This is a mobile-app-augmented, group-delivered version of the six-session Cognitive-Behavioral Treatment for Insomnia that has been disseminated throughout the VA. It incorporates psychoeducation, diary-based sleep assessment, estimation of sleep scheduling and efficiency, evaluation/mitigation of dysfunctional sleep-related beliefs/ behaviors, generation of sleep prescription (typically restriction), iterative review of sleep efficiency and prescription, and planning for maintenance of gains. The mobile-app augmentation substitutes a smartphone-based sleep diary with time-stamping of records to mitigate the common postponement of diary recording and consequent loss of validity. The app also records the sleep prescription, making it, along with links to web-based psychoeducational materials, easily accessible to users. The app also provides plots of bed times, wake times, and sleep efficiency over time, with the goal of promoting adherence.
  Other Names: CBT-I-MA
  Arms: CBT-I-MA
Behavioral: Desensitization Treatment for Insomnia — This is a group-delivered version of the sham sleep improvement treatment developed by Edinger which purports to "desensitize" the patient to the various aspects of the sleep experience which are presented as distressing.
  Other Names: DTI
  Arms: PC

SUMMARY:
The purpose of this study is to investigate the efficacy of a group-based behavioral sleep intervention, and the incremental benefit provided by an adjunct sleep mobile app, on cannabis and sleep outcomes among cannabis dependent Veterans.

DETAILED DESCRIPTION:
The Prevalence of cannabis use disorder (CUD) has been steadily increasing within the Veteran Health Administration (VHA), along with the related significant physical, cognitive, and psychological sequelae. Even in patients with a strong motivation to quit and the presence of empirically-supported interventions, Veterans who receive treatment for CUD have high rates of lapse (63% by 6-months post-treatment) and relapse (71% within 6-months post-treatment). Thus, identifying strategies to improve response to CUD treatment is in the interest of all VHA stakeholders.

Disturbed sleep is common among individuals with CUD and has been shown to result in increased rates of lapse/relapse to cannabis. Providing a behavioral sleep intervention within the context of CUD treatment, and prior to a cessation attempt, has the potential to improve these cessation outcomes.

Cognitive behavioral therapy for insomnia (CBT-I) is a well-established first-line treatment for insomnia. While CBT-I is being disseminated throughout VHA, it is rarely received by Veterans with substance use disorders (SUDs) and, among those that do receive it, it is almost always delivered following a cessation attempt. While CBT-I has been shown to be an effective treatment for improving sleep among individuals with insomnia and co-occurring conditions, including SUDs, there has yet to be an investigation of the impact of providing CBT-I prior to CUD treatment with the goal of improving cessation outcomes. In addition, the development of an adjunct behavioral intervention delivered via mobile app technology within VA holds great promise to bolster outcomes.

The current study seeks to fill this gap by conducting a randomized prospective study designed to evaluate the efficacy of CBT-I, as well as the incremental benefit of including an adjunct sleep mobile app (CBT-I-MA), on both cannabis and sleep outcomes among Veterans with CUD.

ELIGIBILITY:
Inclusion Criteria:

To be included in the current study individuals must

* be a Veteran 18 years or older
* meet Diagnostic and Statistical Manual of Mental Disorders-5 diagnostic criteria for cannabis use disorder;
* meet Diagnostic and Statistical Manual of Mental Disorders diagnostic criteria for insomnia;

Exclusion Criteria:

Individuals will be excluded based on evidence of the following:

* inability to provide fully-informed written consent to participate;
* history of, or current, psychotic symptoms;
* current pregnancy;
* Sleep apnea (>5 on the STOP-Bang assessment);
* active suicidal/homicidal intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Babson, PhD MA BS, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CBT-I-MA: Group Cognitive-Behavioral Therapy for Insomnia Plus Mobile App (CBT-I-MA)
  Cognitive Behavioral Therapy for Insomnia Plus Mobile App (CBT-I-MA): This is a mobile-app-augmented, group-delivered version of the six-session Cognitive-Behavioral Treatment for Insomnia that has been disseminated throughout the VA. It incorporates psychoeducation, diary-based sleep assessment, estimation of sleep scheduling and efficiency, evaluation/mitigation of dysfunctional sleep-related beliefs/behaviors, generation of sleep prescription, iterative review of sleep efficiency and prescription, and planning for maintenance of gains. The mobile-app augmentation substitutes a smartphone-based sleep diary with time-stamping of records to mitigate the common postponement of diary recording and consequent loss of validity. The app also records the sleep prescription, making it easily accessible to users. The app also provides plots of bed times, wake times, and sleep efficiency over time.
- Placebo Control (PC): Desensitization Treatment for Insomnia (DTI)
  Desensitization Treatment for Insomnia: This is a group-delivered version of the sham sleep improvement treatment developed by Edinger which purports to "desensitize" the patient to the various aspects of the sleep experience which are presented as distressing.
Period: Overall Study
Arm/Group | CBT-I | CBT-I-MA | Placebo Control (PC)
Started | 42 | 28 | 41
Completed | 25 | 11 | 24
Not Completed | 17 | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- CBT-I-MA: Group Cognitive-Behavioral Therapy for Insomnia Plus Mobile App (CBT-I-MA)
  Cognitive Behavioral Therapy for Insomnia Plus Mobile App (CBT-I-MA): This is a mobile-app-augmented, group-delivered version of the six-session Cognitive-Behavioral Treatment for Insomnia that has been disseminated throughout the VA. It incorporates psychoeducation, diary-based sleep assessment, estimation of sleep scheduling and efficiency, generation of sleep prescription (typically restriction), iterative review of sleep efficiency and prescription, and planning for maintenance of gains. The mobile-app augmentation substitutes a smartphone-based sleep diary with time-stamping of records to mitigate the common postponement of diary recording and consequent loss of validity. The app also records the sleep prescription, making it, along with links to web-based psychoeducational materials, easily accessible to users.
- Placebo: Desensitization Treatment for Insomnia (DTI)
  Desensitization Treatment for Insomnia: This is a group-delivered version of the sham sleep improvement treatment developed by Edinger which purports to "desensitize" the patient to the various aspects of the sleep experience which are presented as distressing.
- Total: Total of all reporting groups
Arm/Group | CBT-I | CBT-I-MA | Placebo | Total
Number analyzed (Participants) | 25 | 11 | 24 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 11 | 24 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not obtained from one subject.
  years
    number analyzed (Participants) | 24 | 11 | 24 | 59
    (all) | 46.08 (17.49) | 44.27 (13.24) | 52.46 (14.79) | 48.34 (15.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 24 | 10 | 23 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 6
  Not Hispanic or Latino | 20 | 9 | 20 | 49
  Unknown or Not Reported | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 6 | 12
  White | 17 | 6 | 14 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 11 | 24 | 60
marijuana use episodes per week [Mean (Standard Deviation); unit: uses/week] | 12.0051 (12.04773) | 8.0583 (7.59805) | 9.5079 (13.31989) | 10.3 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cannabis Use Frequency Over Time
Description: Measures will include the Timeline Followback for cannabis. All of these measures are standard 7-day point prevalence estimates. In other words, the baseline measure is the number of uses in the 7 days prior to the baseline assessment day. The 6-weeks post-baseline is the number of uses in the 7 days prior to the 6-weeks post-baseline day, and so on.
Time Frame: baseline, 6-weeks post-baseline, 2-weeks post-quit, 4 weeks post-quit, 6-months post-quit
Population: Veteran Cannabis Users
Measure: Mean (Standard Deviation); unit: mean uses per period
Groups:
- CBT-I-MA: Group Cognitive-Behavioral Therapy for Insomnia Plus Mobile App (CBT-I-MA)
  Cognitive Behavioral Therapy for Insomnia Plus Mobile App (CBT-I-MA): This is a mobile-app-augmented, group-delivered version of the six-session Cognitive-Behavioral Treatment for Insomnia that has been disseminated throughout the VA. It incorporates psychoeducation, diary-based sleep assessment, estimation of sleep scheduling and efficiency, evaluation/mitigation of dysfunctional sleep-related beliefs/ behaviors, generation of sleep prescription (typically restriction), iterative review of sleep efficiency and prescription, and planning for maintenance of gains. The mobile-app augmentation substitutes a smartphone-based sleep diary with time-stamping of records to mitigate the common postponement of diary recording and consequent loss of validity. The app also records the sleep prescription, making it, along with links to web-based psychoeducational materials, easily accessible to users.
Arm/Group | CBT-I | CBT-I-MA | Placebo
Number analyzed (Participants) | 25 | 11 | 24
mean uses per period
  baseline | 12.0051 (12.04773) | 8.0583 (7.59805) | 9.5079 (13.31989)
  6-weeks post-baseline: number analyzed (Participants) | 14 | 4 | 16
  6-weeks post-baseline | 11.5714 (13.11763) | 12.6071 (7.58119) | 19.6339 (49.16600)
  2-weeks post-quit: number analyzed (Participants) | 13 | 3 | 14
  2-weeks post-quit | 12.9176 (17.13794) | 10.0476 (6.30247) | 7.5663 (11.02617)
  4 weeks post-quit: number analyzed (Participants) | 12 | 3 | 14
  4 weeks post-quit | 13.6964 (19.53661) | 11.3810 (7.42628) | 4.9388 (4.71061)
  6-months post-quit: number analyzed (Participants) | 9 | 2 | 9
  6-months post-quit | 14.1378 (22.69275) | 17.0000 (4.24264) | 8.7385 (9.77943)

2. Primary Outcome: Point Prevalence Abstinence Over the Three Post-quit Attempt Assessments
Description: point prevalence abstinence will be assessed using the Timeline Follow-back measure for cannabis count of number abstinent
Time Frame: 2-weeks post-quit, 4 weeks post-quit, 6-months post-quit
Population: All participants were considered analyzed by the intent to treat principle, but less than the overall number analyzed contributed data in all three arms. One Placebo participant missing at week 2 rejoined at week 4 and week 6.
Measure: Count of Participants; unit: Participants
Arm/Group | CBT-I | CBT-I-MA | Placebo
Number analyzed (Participants) | 25 | 11 | 24
Participants
  number abstinent at 2 weeks post tx: number analyzed (Participants) | 12 | 3 | 11
  number abstinent at 2 weeks post tx | 0 | 0 | 0
  number abstinent at 4 weeks post tx: number analyzed (Participants) | 11 | 3 | 12
  number abstinent at 4 weeks post tx | 0 | 0 | 0
  number abstinent at 6 months: number analyzed (Participants) | 11 | 3 | 12
  number abstinent at 6 months | 0 | 0 | 0

3. Primary Outcome: Change in Self-reported Sleep Quality Over Time
Description: Self-reported sleep quality will be measured using the Consensus Sleep Diary
Time Frame: 2-weeks post-quit, 4-weeks post-quit, 6-months post-quit
Measure: Count of Participants; unit: Participants
Arm/Group | CBT-I | CBT-I-MA | Placebo
Number analyzed (Participants) | 25 | 11 | 24
Participants | NA — PI is no longer available and project staff could not reconstruct the data and perform the necessary analyses in a manner that would yield valid results. | NA — PI is no longer available and project staff could not reconstruct the data and perform the necessary analyses in a manner that would yield valid results. | NA — PI is no longer available and project staff could not reconstruct the data and perform the necessary analyses in a manner that would yield valid results.

4. Primary Outcome: Change in Objective Sleep Quality Over Time
Description: Objective sleep quality will be measured via actigraphy
Time Frame: 2-weeks post-quit, 4-weeks post-quit, 6-months post-quit
Measure: Count of Participants; unit: Participants
Arm/Group | CBT-I | CBT-I-MA | Placebo
Number analyzed (Participants) | 25 | 11 | 24
Participants | NA — PI is no longer available and project staff could not reconstruct the data and perform the necessary analyses in a manner that would yield valid results. | NA — PI is no longer available and project staff could not reconstruct the data and perform the necessary analyses in a manner that would yield valid results. | NA — PI is no longer available and project staff could not reconstruct the data and perform the necessary analyses in a manner that would yield valid results.

ADVERSE EVENTS:
Time Frame: Duration of study participation - 6 weeks of tx + 6 months safety f/u
Description: No difference
Arm/Group | CBT-I | CBT-I-MA | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/11 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/11 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/11 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-02-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT02102230/SAP_000.pdf
  • Study Protocol (2015-06-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT02102230/Prot_001.pdf